CLINICAL TRIAL: NCT05099068
Title: A Prospective Longitudinal Profiling Program of Cancer Patients With Sequential Tumor and Liquid Biopsies
Brief Title: Profiling Program of Cancer Patients With Sequential Tumor and Liquid Biopsies (PLANET)
Acronym: PLANET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Plasticity Longitudinal cANcer
Record Dates: First submitted 2021-07-30; First posted 2021-10-29 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Advanced / Metastic Solid Tumors; Glioblastoma; Chronic Leukemia Lymphocytic
Keywords: Molecular Screening; Genomic profiles; Transcriptomic profiles
MeSH Terms: conditions — Glioblastoma; Leukemia, B-Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IMMUNOTHERAPY COHORTS (Experimental): This cohort include following cancers treated with immunotherapy : metastatic Small cell lung cancer (SLCC); recurrent/Metastatic Head and Neck squamous cell carcinoma (HNSCC); MSI-High, any tumor types and HPV-related cancers,any tumor types
  Interventions: Biological: Blood and tumor samples
- TARGETED THERAPIES COHORTS (Experimental): This cohort include following cancers treated with targeted therapies : Metastatic GIST; BRAF-mutated tumors (CRC (BRAF V600E), lung (V600 only) and thyroid (all BRAF mutation with known sensitivity to Dabrafenib) cancer); All solid tumor types with RET fusion / mutation and Chronic Lymphocytic Leukemia (CLL) in the relapsed setting.
  Interventions: Biological: Blood and tumor samples
- CHEMOTHERAPY COHORTS (Experimental): This cohort include following cancers treated with chemotherapies : metastatic Small cell lung cancer (SLCC); recurrent/Metastatic Head and Neck squamous cell carcinoma (HNSCC); Metastatic Triple negative breast cancer (TNBC); Glioblastoma; Advanced high grade epithelial ovarian cancer
  Interventions: Biological: Blood and tumor samples

INTERVENTIONS:
Biological: Blood and tumor samples — Longitudinal molecular profiling of tumor and liquid biopsies.

SUMMARY:
The proposal is to conduct a prospective, multi-cohort study aiming to decipher molecular profiles/biological characteristics of advanced cancer patients during the course of their disease with longitudinal and sequential analyses of tumor and liquid biopsies. This approach will allow i) to develop a model in order to predict tumor response / resistance in real life conditions and to better understand adaptive mechanisms and ii) to potentially propose therapeutic options to enrolled patients following the review of the biological/molecular data generated during this study and during a Molecular Tumor Board in case of disease progression. This study will include 12 cohorts according to tumor type and standard treatment received (See Inclusion criteria I1). Patient will be enrolled before the initiation of standard anti-cancer treatment.

DETAILED DESCRIPTION:
Most of the molecular screening programs have allowed to successfully guide patients to personalized therapy only for a minority of patients (10-20%) and few patients have actually benefit from these programs with low objective response under personalized therapy.

During the course of disease and / or of treatment, tumors become more heterogeneous and include a collection of cells harboring distinct molecular signatures with differential levels of sensitivity to treatment. Assessment of tumor heterogeneity and plasticity are essential for the development of effective therapies. Longitudinal analysis of biopsy samples is of considerable interest to assess the complex clonal architecture of cancers and potentially adapt cancer treatment to tumor profile/characteristics overtime. In this context, profiling of circulating tumor DNA using non-invasive liquid biopsies is also an interesting approach to assess cancer evolution by showing the contribution of clonal heterogeneity to chemotherapy resistance and metastasis in high-risk patients.

The proposal is to conduct a prospective, multi-cohort study aiming to decipher molecular profiles/biological characteristics of advanced cancer patients during the course of their disease with longitudinal and sequential analyses of tumor and liquid biopsies. This approach will allow i) to develop a model in order to predict tumor response / resistance in real life conditions and to better understand adaptive mechanisms and ii) to potentially propose therapeutic options to enrolled patients following the review of the biological/molecular data generated during this study and during a Molecular Tumor Board in case of disease progression. This study will include 12 cohorts according to tumor type and standard treatment received (See Inclusion criteria I1). Patient will be enrolled before the initiation of standard anti-cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

I1. Adult male or female patient with confirmed diagnosis of advanced/metastatic cancer to be treated with standard anti-cancer treatment according to :

* For metastatic Small cell lung cancer (SLCC) : treatment by Immunotherapy ± chemotherapy
* For Recurrent/Metastatic Head and Neck squamous cell carcinoma (HNSCC) : treatment by Immunotherapy (all lines) ± chemotherapy if in agreement with SmPC
* For Metastatic Urothelial carcinoma : treatment by 1st line chemotherapy with avelumab as maintenance treatment (patients will be enrolled following 4 to 6 cycles of CT, only patient initiating avelumab maintenance are eligible (i.e. patients with SD or PR after CT)
* For MSI-High, any tumor types : treatment by Immunotherapy
* For HPV-related cancers, any tumor types : treatment by Immunotherapy
* Metastatic GIST : treatment by Imatinib
* BRAF- V600E tumors (lung and thyroid cancer) : treatment by Dabrafenib + trametinib
* BRAF- mutated tumors (CRC, lung and thyroid cancer) :

Lung (V600E only) and thyroid (all BRAF mutation with known sensitivity to Dabrafenib): treatment by Dabrafenib + trametinib CRC (BRAF V600E): treatment by Encorafenib + cetuximab

* All solid tumor types with ret fusion / mutation : treatment by Selpercatinib
* Metastatic Triple negative breast cancer (TNBC) : treatment by 1st line chemotherapy
* Glioblastoma : treatment by Radiochemotherapy
* Advanced high grade epithelial ovarian cancer : treatment by 1st line Chemotherapy
* Chronic Lymphocytic Leukemia (CLL) in the relapsed setting : treatment by Bruton Kinase Inhibitors

I2. All solid tumor cohorts: Availability of an archival representative formalin-fixed paraffin-embedded (FFPE) tumor sample [...]

I3. All solid tumor cohorts: Disease evaluable as per RECIST V1.1

I4. All solid tumor cohorts excluding Glioblastoma: Tumor lesion visible by medical imaging and accessible to repeatable percutaneous or endoscopic mandatory de novo tumor sampling [...]

I5. Performance status (PS) ECOG 0 or 1.

I6. Patient should understand, sign, and date the written ICF prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures including sequential tumor biopsies as per protocol.

I7. Patient must be covered by a medical insurance.

Exclusion Criteria:

NI1. All solid tumor cohorts - Patient with non-acceptable tumor sample at screening.

NI2. Any condition contraindicated with blood/tumor sampling procedures required by the protocol.

NI3. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.

NI4. Pregnant or breast-feeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients with meaningful molecular genetic alterations on tumor sample | At the end of study (4 years)
  Identification of molecular genetic alterations based on molecular characterisation (WES and RNASeq) of tumor at diagnosis, then under standard anti-cancer treatment : treatment start, 1st radiological evaluation and disease progression
Number of patients with meaningful molecular genetic alterations on circulating tumour DNA (ctDNA) | At the end of study (4 years)
  Identification of molecular genetic alterations based on molecular characterisation (WES and RNASeq) of ctDNA under standard anti-cancer treatment : treatment start, each radiological evaluation and disease progression
Number of patients with meaningful immunological features | At the end of study (4 years)
  Identification and characterisation of the tumor microenvironment and the host's immunological profile, at diagnosis and during patient treatment
Objective Response Rate (ORR) as per RECIST V1.1 and according to central review | 3 months
  For solid tumors excluding glioblastoma only
Progression-Free Survival (PFS) | 6 months
  For glioblastoma only
Objective Response Rate (ORR) according to iwCLL criteria | 6 months
  For chronic lymphocytic leukemia

SECONDARY OUTCOMES:
Correlation between disease evolution and molecular and/or immunological biomarkers | Time Frame: up to 4 years
  To identify potential prognostic and predictive biomarkers on tumor samples collected during patient's treatment and follow-up detected by molecular biology techniques, and on immunological findings
Evaluation of circulating-tumor DNA (ctDNA; liquid biopsy) yields similar genomic profile as the tumor sample. | 48 months
  To identify potential prognostic and predictive biomarkers based on changes on circulating tumour DNA (ctDNA), detected by molecular biology techniques
Number of patients with recommended therapy according to biological data (liquid versus tumor biopsy) | 48 months
Tumor characteristics using a radiomic approach and detailed analyses of imaging. | 48 months
FACT-G questionnaire | 48 months
  To evaluate the quality of life and emotional distress anxiety/depression over time of patients
HADS questionnaire | 48 months
  To evaluate the quality of life and emotional distress anxiety/depression over time of patients
PRO questionnaire | 48 months
  To evaluate the quality of life and emotional distress anxiety/depression over time of patients
Correlation between patient's understanding and experiences of precision medicine clinical trial | 48 months
  Measured by thematic analysis of semi-structured interviews: themes and sub-themes will be analyzed in order to develop items for the construction and validation of a quantitative questionnaire.
Correlation between socio-spatial inequalities in access to the PLANET program and the impact on the quality of life of patients | 48 months
  Questionnaire
TKI pharmacokinetics | 48 months
  Plasma concentrations of TKI

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SAINTIGNY, MD, PhD, Principal Investigator — Centre Leon Berard
Locations (2):
- France (2):
  - HOPITAL Pierre WERTHEIMER - HCL, Bron
  - Centre Léon Bérard, Lyon